CLINICAL TRIAL: NCT01122264
Title: Impact of Tadalafil (LY450190) Once a Day or Tadalafil on Demand Compared to Sildenafil Citrate on Demand on Treatment Discontinuation in Patients With Erectile Dysfunction Who Are naïve to PDE5 Inhibitors
Brief Title: A Study in Patients With Erectile Dysfunction
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 13085; H6D-EW-LVIJ (Other: Eli Lilly and Company)
Record Dates: First submitted 2010-05-05; First posted 2010-05-13 (Estimated); Results first posted 2012-10-19 (Estimated); Last update posted 2012-10-19 (Estimated); Status verified 2012-09

CONDITIONS: Erectile Dysfunction
Keywords: Erectile Dysfunction
MeSH Terms: conditions — Erectile Dysfunction | interventions — Tadalafil; Sildenafil Citrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Tadalafil on demand (Experimental): 10 milligrams (mg) or 20 mg on demand
  Interventions: Drug: Tadalafil
- Tadalafil once a day (Experimental): 5 mg or 2.5 mg once a day
  Interventions: Drug: Tadalafil
- Sildenafil Citrate (Active Comparator): 50 mg, 100 mg, or 25 mg on demand
  Interventions: Drug: Sildenafil Citrate

INTERVENTIONS:
Drug: Tadalafil — Administered orally for 24 weeks.
  Other Names: Cialis; LY450190
  Arms: Tadalafil on demand; Tadalafil once a day
Drug: Sildenafil Citrate — Administered orally for 24 weeks.
  Arms: Sildenafil Citrate

SUMMARY:
The purpose of this study is to investigate if treatment in erectile dysfunction with a long-acting drug (Tadalafil) taken once a day or taken as needed results in a longer treatment adherence and better long term outcomes (over 24 weeks), compared with a short-acting drug (Sildenafil Citrate) taken as needed.

ELIGIBILITY:
Inclusion Criteria:

* History of Erectile Dysfunction (ED) of at least 3 months duration.
* Anticipate having the same adult female sexual partner during the study.
* Agree not to use any other treatment for ED and to participate in recording responses to questionnaires and other instruments used in this study.

Exclusion Criteria:

* Previous or current treatment with tadalafil or any other phosphodiesterase type 5 (PDE5) inhibitor.
* ED caused by other primary sexual disorders, history of radical prostatectomy or other pelvic surgery with subsequent failure to achieve any erection, or history of penile implant or clinically significant penile deformity.
* ED caused by untreated or inadequately treated endocrine disease.
* Current treatment with doxazosin, nitrates, cancer chemotherapy, or anti-androgens.
* Severe renal or hepatic impairment, history of malignant hypertension.
* Presence or history of specific heart conditions.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 770 (Actual)
Dates: Start 2010-05; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (45):
- France (11):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Carpentras
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chambéry
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., La Bouëxière
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lyon
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marseille
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Montpellier
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mûrs-Erigné
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Nantes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rennes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Toulouse
- Germany (10):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Giengen an der Brenz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Grevenbroich
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Holzminden
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Koblenz
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leipzig
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Leverkusen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lübeck
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Marburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Mühlacker
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warburg
- Greece (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Heraklion
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Larissa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Pátrai
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Thessaloniki
- Poland (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Kutno
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Legionowo
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Warsaw
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wroclaw
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Porto, Portugal
- Romania (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bucharest
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cluj-Napoca
- Spain (9):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alcorcón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aravaca
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Coslada
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Gijón
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Málaga
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., San Sebastián de los Reyes
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Vigo
- United Kingdom (3):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Fowey, Cornwall
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Durham, County Durham
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Plymouth, Devon

REFERENCES:
- [Derived] Buvat J, Buttner H, Hatzimouratidis K, Vendeira PA, Moncada I, Boehmer M, Henneges C, Boess FG. Adherence to initial PDE-5 inhibitor treatment: randomized open-label study comparing tadalafil once a day, tadalafil on demand, and sildenafil on demand in patients with erectile dysfunction. J Sex Med. 2013 Jun;10(6):1592-602. doi: 10.1111/jsm.12130. Epub 2013 Apr 2. PMID 23551622

RESULTS

PARTICIPANT FLOW:
Groups:
- Tadalafil On Demand: Participants were instructed to take a 10-milligram (mg) or 20-mg tablet of tadalafil orally on demand, with a maximum of 4 tablets per week (and no more than 1 tablet per day) for 24 weeks.
- Tadalafil Once a Day: Participants were instructed to take a 5-mg or 2.5-mg tablet of tadalafil orally once a day for 24 weeks.
- Sildenafil Citrate On Demand: Participants were instructed to take a 50-mg, 100-mg, or 25-mg tablet of sildenafil citrate orally on demand, with a maximum of 4 tablets per week (and no more than 1 tablet per day) for 24 weeks.
Period: Overall Study
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Started | 252 | 257 | 261
Received at Least 1 Dose of Study Drug | 250 | 257 | 260
Completed | 220 | 228 | 214
Not Completed | 32 | 29 | 47
Not completed — Adverse Event | 6 | 5 | 7
Not completed — Death | 1 | 0 | 0
Not completed — Lost to Follow-up | 5 | 9 | 13
Not completed — Entry Criteria Not Met | 1 | 0 | 0
Not completed — Protocol Violation | 7 | 7 | 9
Not completed — Withdrawal by Subject | 6 | 6 | 16
Not completed — Physician Decision | 3 | 1 | 1
Not completed — Lack of Efficacy | 3 | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand | Total
Number analyzed (Participants) | 252 | 257 | 261 | 770
Age Continuous [Mean (Standard Deviation); unit: years] | 53.2 (11.57) | 52.9 (11.69) | 53.0 (11.76) | 53.0 (11.66)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 252 | 257 | 261 | 770
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 4 | 4 | 10
  White | 248 | 251 | 254 | 753
  More than one race | 0 | 0 | 1 | 1
  Unknown or Not Reported | 2 | 2 | 2 | 6
Region of Enrollment [Number; unit: participants]
  Portugal | 6 | 5 | 7 | 18
  France | 99 | 102 | 100 | 301
  Greece | 9 | 8 | 9 | 26
  Poland | 15 | 16 | 16 | 47
  Spain | 48 | 49 | 52 | 149
  Romania | 20 | 22 | 21 | 63
  Germany | 45 | 45 | 47 | 137
  United Kingdom | 10 | 10 | 9 | 29

OUTCOME MEASURES:

1. Primary Outcome: Time to Discontinuation of Randomized Treatment
Description: Time to discontinuation of randomized treatment was defined as the number of days from randomization until the day the participant discontinued the randomized treatment. Discontinuation of randomized treatment was defined as switching between the 3 study treatments (tadalafil on demand, tadalafil once a day, or sildenafil citrate on demand) or discontinuing from all treatments. A change of dose within the same treatment was not considered switching of treatment. This outcome measure was estimated using the Kaplan-Meier product-limit method.
Time Frame: Baseline up to 334 days
Population: The analysis included all randomly assigned participants.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 252 | 257 | 261
days | NA [187 to NA] — The median and the 95% confidence interval were not estimable because an insufficient number of participants reached the event at the time of the data cutoff. | 130 [113 to NA] — The 95% confidence interval was not estimable because an insufficient number of participants reached the event at the time of the data cutoff. | 67 [64 to 77]
Statistical Analysis 1: Comparison: Tadalafil Once a Day vs Sildenafil Citrate On Demand; Test type: Superiority or Other; p < 0.001, Regression, Cox — P-value: Tadalafil Once a Day versus Sildenafil Citrate On Demand treatment groups. Cox's proportional hazards model with factors for randomized treatment group, baseline International Index of Erectile Function-Erectile Function score, and country; Cox Proportional Hazard = 0.66, 97.3% CI 2-sided [0.51 to 0.85]
Statistical Analysis 2: Comparison: Tadalafil On Demand vs Sildenafil Citrate On Demand; Test type: Superiority or Other; p < 0.001, Regression, Cox — P-value: Tadalafil On Demand versus Sildenafil Citrate On Demand treatment groups. Cox's proportional hazards model with factors for randomized treatment group, baseline International Index of Erectile Function-Erectile Function score, and country; Cox Proportional Hazard = 0.49, 97.3% CI 2-sided [0.37 to 0.65]
Statistical Analysis 3: Comparison: Tadalafil On Demand vs Tadalafil Once a Day; Test type: Superiority or Other; p = 0.033, Regression, Cox — P-value: Tadalafil On Demand versus Tadalafil Once a Day treatment groups using Cox's proportional hazards model with factors for randomized treatment group, baseline International Index of Erectile Function-Erectile Function score, and country; Cox Proportional Hazard = 1.32, 95% CI 2-sided [1.02 to 1.71]

2. Secondary Outcome: Change From Baseline to 4, 8, 16 and 24 Weeks of the International Index of Erectile Function (IIEF) Erectile Function (EF) Domain
Description: Self-reported EF score over past 4 weeks. Items 1-5 scores range from 0 (no sexual activity) to 5 (high EF). Item 15 score ranges from 1 (very low confidence to get/keep erection) to 5 (very high confidence). Total scores range from 1 to 30; lower scores denote greater erectile dysfunction severity. Least Squares Mean changes from baseline to endpoint for each visit from repeated measures analysis included terms for baseline score, treatment group, country, baseline*treatment (if p<0.10), visit, and visit*treatment. Correlation matrix for repeated observations assumed to be unstructured.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline IIEF-EF observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 241 | 251 | 250
units on a scale
  Change from Baseline to Week 4 | 7.92 (0.44) | 8.60 (0.43) | 8.86 (0.43)
  Change from Baseline to Week 8 (n=231, 232, 232) | 8.98 (0.45) | 9.08 (0.45) | 9.70 (0.44)
  Change from Baseline to Week 16 (n=167, 146, 101) | 10.60 (0.41) | 9.93 (0.42) | 10.56 (0.45)
  Change from Baseline to Week 24 (n=141, 116, 81) | 10.70 (0.43) | 10.01 (0.45) | 11.05 (0.49)

3. Secondary Outcome: Change From Baseline to 4, 8, 16 and 24 Weeks of the International Index of Erectile Function (IIEF) Orgasmic Function Domain
Description: Self-reported orgasmic function on the IIEF over past 4 weeks and consists of 2 questions (items 9 and 10). Each question is rated on a scale from 0 (no sexual stimulation) to 5 (almost always/always). Total scores range from 0 to 10; lower scores represent lower orgasmic function. Least Squares Mean changes from baseline to endpoint for each visit were from a repeated measures analysis and included terms for baseline score, treatment group, country, baseline*treatment (if p<0.10), visit, and visit*treatment. The correlation matrix for the repeated observations was assumed to be unstructured.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline IIEF Orgasmic Function observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 241 | 251 | 250
units on a scale
  Change from Baseline to Week 4 | 1.64 (0.16) | 1.75 (0.16) | 1.92 (0.16)
  Change from Baseline to Week 8 (n=231, 232, 232) | 1.77 (0.16) | 2.08 (0.16) | 2.26 (0.16)
  Change from Baseline to Week 16 (n=167, 146, 101) | 2.37 (0.15) | 2.25 (0.16) | 2.66 (0.17)
  Change from Baseline to Week 24 (n=141, 116, 81) | 2.55 (0.15) | 2.48 (0.16) | 2.62 (0.18)

4. Secondary Outcome: Change From Baseline to 4, 8, 16 and 24 Weeks of the International Index of Erectile Function (IIEF) Sexual Desire Domain
Description: Self-reported sexual desire on IIEF over past 4 weeks; comprises 2 questions (items 11 and 12). Each question rated on a scale from 1 (almost never or low/no sexual desire) to 5 (almost always or very high sexual desire). Total scores range: 2 to 10; lower numerical scores denote lower sexual desire. Least Squares Mean changes from baseline to endpoint for each visit from repeated measures analysis and included terms for baseline score, treatment group, country, baseline*treatment (if p<0.10), visit, and visit*treatment. Correlation matrix for repeated observations assumed to be unstructured.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline IIEF Sexual Desire observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 244 | 250 | 249
units on a scale
  Change from Baseline to 4 Weeks | 0.77 (0.10) | 0.75 (0.10) | 0.69 (0.10)
  Change from Baseline to 8 Weeks (n=230, 232, 232) | 0.96 (0.11) | 0.90 (0.11) | 0.87 (0.11)
  Change from Baseline to 16 Weeks (n=167, 146, 101) | 1.15 (0.12) | 0.87 (0.12) | 1.07 (0.14)
  Change from Baseline to 24 Weeks (n=140, 117, 81) | 1.19 (0.12) | 0.78 (0.13) | 1.29 (0.14)

5. Secondary Outcome: Change From Baseline to 4, 8, 16 and 24 Weeks of the Sexual Encounter Profile (SEP)
Description: Participant-assessed diary. Has 5 questions (Question[Q]1:erection achievement, Q2:successful penetration, Q3:successful intercourse, Q4:satisfied with erection, and Q5:satisfied with sexual experience) for each sexual encounter made over specified period of time. SEP Q1-Q5 scores determined as percentage of 'Yes' responses to each of 5 questions out of all sexual attempts recorded during the time period. Least Squares Mean changes from baseline to endpoint for each visit from a repeated measures analysis included terms for baseline score, treatment group, country, visit, and visit*treatment.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline SEP observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of "yes" responses
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 242 | 246 | 248
percentage of "yes" responses
  Q1:Change from Baseline to 4 Weeks | 14.50 [11.82 to 17.18] | 18.49 [15.83 to 21.14] | 18.41 [15.77 to 21.05]
  Q1:Change from Baseline to 8 Weeks (n=224,231,229) | 16.62 [14.05 to 19.19] | 19.88 [17.33 to 22.43] | 20.41 [17.87 to 22.96]
  Q1:Change from Baseline to 16 Weeks (n=166,146,99) | 18.46 [16.02 to 20.89] | 19.19 [16.72 to 21.67] | 20.58 [17.90 to 23.27]
  Q1:Change from Baseline to 24 Weeks (n=139,115,81) | 19.97 [17.78 to 22.15] | 19.60 [17.33 to 21.86] | 20.34 [17.94 to 22.74]
  Q2:Change from Baseline to 4 Weeks | 27.48 [23.77 to 31.19] | 28.56 [24.87 to 32.24] | 29.64 [25.96 to 33.31]
  Q2:Change from Baseline to 8 Weeks (n=224,231,229) | 31.16 [27.57 to 34.76] | 31.66 [28.09 to 35.22] | 34.08 [30.52 to 37.64]
  Q2:Change from Baseline to 16 Weeks (n=166,146,99) | 32.76 [29.38 to 36.14] | 32.76 [29.33 to 36.20] | 36.07 [32.38 to 39.76]
  Q2:Change from Baseline to 24 Weeks (n=139,115,81) | 35.83 [32.71 to 38.94] | 34.70 [31.48 to 37.92] | 35.93 [32.51 to 39.35]
  Q3:Change from Baseline to 4 Weeks | 41.52 [36.79 to 46.26] | 41.76 [37.05 to 46.47] | 44.45 [39.76 to 49.13]
  Q3:Change from Baseline to 8 Weeks (n=224,231,229) | 47.45 [42.65 to 52.26] | 44.58 [39.80 to 49.35] | 52.11 [47.36 to 56.86]
  Q3:Change from Baseline to 16 Weeks (n=166,146,99) | 54.26 [49.86 to 58.67] | 50.62 [46.14 to 55.11] | 56.96 [52.10 to 61.82]
  Q3:Change from Baseline to 24 Weeks (n=139,115,81) | 56.39 [51.89 to 60.89] | 53.83 [49.13 to 58.53] | 56.28 [51.18 to 61.38]
  Q4:Change from Baseline to 4 Weeks | 49.59 [44.22 to 54.97] | 51.78 [46.44 to 57.12] | 51.45 [46.13 to 56.76]
  Q4:Change from Baseline to 8 Weeks (n=224,231,229) | 60.86 [55.37 to 66.36] | 55.59 [50.14 to 61.05] | 59.28 [53.85 to 64.71]
  Q4:Change from Baseline to 16 Weeks (n=166,146,99) | 66.17 [60.92 to 71.43] | 63.00 [57.64 to 68.36] | 66.48 [60.65 to 72.31]
  Q4:Change from Baseline to 24 Weeks (n=139,115,81) | 72.67 [67.46 to 77.89] | 68.06 [62.58 to 73.54] | 69.04 [63.06 to 75.02]
  Q5:Change from Baseline to 4 Weeks | 46.12 [40.79 to 51.46] | 45.71 [40.41 to 51.01] | 49.63 [44.35 to 54.90]
  Q5:Change from Baseline to 8 Weeks (n=224,231,229) | 53.92 [48.46 to 59.37] | 50.06 [44.65 to 55.47] | 55.73 [50.33 to 61.13]
  Q5:Change from Baseline to 16 Weeks (n=166,146,99) | 61.57 [56.26 to 66.88] | 54.56 [49.16 to 59.96] | 62.40 [56.55 to 68.25]
  Q5:Change from Baseline to 24 Weeks (n=139,115,81) | 65.45 [60.29 to 70.60] | 62.17 [56.78 to 67.57] | 66.57 [60.72 to 72.42]

6. Secondary Outcome: Global Assessment Questions (GAQ)
Description: The GAQ consists of 2 Yes/No/No Response (No Respo) questions. GAQ Question (Q)1: Has the treatment you have been taking during this study improved your erections? GAQ Q2: Has the treatment improved your ability to engage in sexual activity?
Time Frame: 24 weeks
Population: The analysis included all randomly assigned participants. The last available GAQ assessment for each participant was used in the analysis.
Measure: Number; unit: participants
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 252 | 257 | 261
participants
  Q1:Treatment improved erections? Yes | 218 | 219 | 203
  Q1:Treatment improved erections? No | 20 | 23 | 34
  Q1: Treatment improved erections? No Response | 14 | 15 | 24
  Q2:Treatment improved ability to engage? Yes | 209 | 214 | 204
  Q2:Treatment improved ability to engage? No | 14 | 7 | 8
  Q2: Treatment improved ability to engage? No Respo | 29 | 36 | 49

7. Secondary Outcome: Number of Treatment Switches
Description: The number of times participants switched erectile dysfunction medication within the 3 treatments being studied (tadalafil on demand, tadalafil once a day, or sildenafil citrate on demand).
Time Frame: Baseline through 24 weeks
Population: The analysis included all randomly assigned participants who switched erectile dysfunction medication and had a baseline and post-baseline observation.
Measure: Mean (Standard Deviation); unit: number of treatment switches
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 87 | 120 | 151
number of treatment switches | 1.2 (0.4) | 1.2 (0.5) | 1.3 (0.5)

8. Secondary Outcome: Patterns of Erectile Dysfunction Treatment Change
Description: Results are reported as the number of participants per sequence of study medications (tadalafil on demand, tadalafil once a day, or sildenafil citrate on demand) that were taken as a result of switching treatments. The Other Treatment Sequence reports the number of participants per sequence of study medications that were taken as a result of switching treatments more than once. The number of participants who did not switch is also reported.
Time Frame: Baseline through 24 weeks
Population: All randomly assigned participants were included in the analysis.
Measure: Number; unit: participants
Groups:
- Entire Study Population: Tadalafil On Demand: Participants were instructed to take a 10-milligram (mg) or 20-mg tablet of tadalafil orally on demand, with a maximum of 4 tablets per week (and no more than 1 tablet per day).
  Tadalafil Once a Day: Participants were instructed to take a 5-mg or 2.5-mg tadalafil tablet orally, once a day.
  Sildenafil Citrate On Demand: Participants were instructed to take a 50-mg, 100-mg, or 25-mg tablet of sildenafil citrate orally on demand, with a maximum of 4 tablets per week (and no more than 1 tablet per day).
Arm/Group | Entire Study Population
Number analyzed (Participants) | 770
participants
  No Treatment Intake | 3
  No Switch | 409
  From Once a Day to Any On Demand | 95
  From Any On Demand to Once a Day | 84
  From Any On Demand to Any On Demand | 97
  Returning Back to Randomized Treatment | 35
  Other Treatment Sequence | 47

9. Secondary Outcome: Reasons for Discontinuation of Randomized Erectile Dysfunction Treatment
Description: The reported reasons for a decision to discontinue from initial randomized treatment prior to Week 24 are reported. Discontinuation of randomized treatment was defined as switching between the 3 study treatments (tadalafil on demand, tadalafil once a day, or sildenafil citrate on demand) or discontinuing from all treatments. A change of dose within the same treatment was not considered as switching of treatment.
Time Frame: Baseline through 24 weeks
Population: The analysis included all randomly assigned participants.
Measure: Number; unit: participants
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 252 | 257 | 261
participants
  Slow onset of action | 5 | 9 | 10
  Completed treatment | 1 | 1 | 1
  Lack of efficacy (hardness of erection) | 46 | 55 | 55
  Lack of efficacy (duration of erection) | 7 | 11 | 24
  Lack of confidence in medication working each time | 3 | 5 | 2
  Adverse event | 7 | 10 | 16
  Feel medication controls my sexual life | 1 | 0 | 7
  Non-desired spontaneous erections | 2 | 4 | 0
  Time constraints due to short drug action window | 1 | 0 | 11
  Partner's request | 0 | 2 | 3
  Don't want to take a pill every day | 0 | 27 | 0
  Prefer a pill every day, not on demand | 20 | 0 | 28
  Participant discontinuation from the trial | 11 | 11 | 14
  Participant did not take any study drug | 2 | 0 | 1
  Participants without discontinuation event | 146 | 122 | 89

10. Secondary Outcome: Number of Days From the 8-Week Study Visit to the Time the Participant Discontinues From All Phosphodiesterase Type 5 (PDE5) Inhibitor Treatments
Description: The differences in time between the 8-week time point and the discontinuation of all study treatments (that is, discontinuation from the study and not switching to another treatment) are reported by the median (95% confidence interval). Duration was measured as the number of days from Week 8 to the date of the last dose of the study drug. This outcome measure was estimated using the Kaplan-Meier product-limit method.
Time Frame: 8 weeks up to 334 days
Population: The analysis included all randomly assigned participants who completed the 8-week randomized treatment.
Measure: Median (95% Confidence Interval); unit: days
Groups:
- Tadalafil On Demand: Participants were instructed to take a 10-milligram (mg) or 20-mg tablet of tadalafil orally on demand, with a maximum of 4 tablets per week (and no more than 1 tablet per day).
- Tadalafil Once a Day: Participants were instructed to take a 5-mg or 2.5-mg tadalafil tablet orally, once a day.
- Sildenafil Citrate On Demand: Participants were instructed to take a 50-mg, 100-mg, or 25-mg tablet of sildenafil citrate orally on demand, with a maximum of 4 tablets per week (and no more than 1 tablet per day).
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 234 | 238 | 236
days | NA [NA to NA] — The median and the 95% confidence interval were not estimable because an insufficient number of participants reached the event at the time of the data cutoff. | NA [200 to NA] — The median and the 95% confidence interval were not estimable because an insufficient number of participants reached the event at the time of the data cutoff. | 187 [165 to NA] — The 95% confidence interval was not estimable because an insufficient number of participants reached the event at the time of the data cutoff.

11. Secondary Outcome: Change From Baseline to 4, 8, 16 and 24 Weeks of the International Index of Erectile Function (IIEF) Intercourse Satisfaction Domain
Description: Self-reported intercourse satisfaction score over past 4 weeks (1 intercourse attempt item, 2 intercourse satisfaction items). Each item range: 0 (no intercourse attempts/no satisfaction) to 5 (more attempts/high satisfaction). Total scores range: 0-15; lower scores=lower intercourse satisfaction. Least Squares Mean changes from baseline to endpoint for each visit from repeated measures analysis and included terms for baseline score, treatment group, country, baseline*treatment (if p<0.10), visit, and visit*treatment. Correlation matrix for repeated observations assumed to be unstructured.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline IIEF Intercourse Satisfaction observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 242 | 251 | 251
units on a scale
  Change from Baseline to Week 4 | 3.21 (0.20) | 3.22 (0.20) | 3.53 (0.20)
  Change from Baseline to Week 8 (n=231, 232, 232) | 3.69 (0.20) | 3.15 (0.20) | 3.95 (0.20)
  Change from Baseline to Week 16 (n=167, 146, 101) | 4.38 (0.20) | 3.60 (0.21) | 4.41 (0.23)
  Change from Baseline to Week 24 (n=141, 116, 81) | 4.48 (0.21) | 3.71 (0.22) | 4.70 (0.24)

12. Secondary Outcome: Change From Baseline to 4, 8, 16 and 24 Weeks of the International Index of Erectile Function (IIEF) Overall Satisfaction Domain
Description: Self-reported overall satisfaction on the IIEF over past 4 weeks and consists of 2 questions (items 13 and 14), each rated on a scale from 1 (very dissatisfied) to 5 (very satisfied). Total scores range from 2 to 10; lower numerical scores represent lower overall satisfaction. Least Squares Mean changes from baseline to endpoint for each visit were from a repeated measures analysis and included terms for baseline score, treatment group, country, baseline*treatment (if p<0.10), visit, and visit*treatment. The correlation matrix for the repeated observations was assumed to be unstructured.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline IIEF Overall Satisfaction observation.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 245 | 250 | 251
units on a scale
  Change from Baseline to Week 4 | 2.46 (0.16) | 2.58 (0.15) | 2.72 (0.15)
  Change from Baseline to Week 8 (n=230, 231, 233) | 2.80 (0.16) | 2.85 (0.16) | 2.98 (0.16)
  Change from Baseline to Week 16 (n=167, 145, 101) | 3.34 (0.15) | 3.09 (0.15) | 3.48 (0.17)
  Change from Baseline to Week 24 (n=141, 116, 81) | 3.50 (0.15) | 3.24 (0.16) | 3.41 (0.17)

13. Secondary Outcome: Erectile Dysfunction Inventory of Treatment Satisfaction (EDITS) Questionnaire at 4, 8, 16, and 24 Weeks
Description: The participant questionnaire consists of 11 questions. Each question is rated on a scale of 0 (extremely low treatment satisfaction) to 4 (extremely high treatment satisfaction). The EDITS summary score was obtained by adding each individual result for all questions, dividing by the number of questions answered (mean satisfaction score), then multiplying by 25, thus obtaining a score range from 0 (extremely low treatment satisfaction) to 100 (extremely high satisfaction). Least Squares Mean changes were adjusted for treatment group, country, visit, and visit*treatment.
Time Frame: 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline EDITS observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 246 | 252 | 249
units on a scale
  EDITS at Week 4 | 72.36 [69.64 to 75.08] | 75.20 [72.51 to 77.90] | 71.98 [69.28 to 74.67]
  EDITS at Week 8 (n=231, 235, 231) | 75.28 [72.51 to 78.05] | 76.64 [73.88 to 79.39] | 72.74 [69.99 to 75.49]
  EDITS at Week 16 (n=168, 147, 100) | 79.64 [77.00 to 82.29] | 77.66 [74.97 to 80.35] | 76.64 [73.71 to 79.56]
  EDITS at Week 24 (n=141, 118, 80) | 81.01 [78.44 to 83.58] | 78.75 [76.10 to 81.41] | 77.98 [75.09 to 80.87]

14. Secondary Outcome: Change From Baseline to 24 Week Endpoint of the Sexual Self-Confidence, Spontaneity, and Time Concerns Domains (23-items) of the Psychological and Interpersonal Relationships Scale (PAIRS)
Description: The PAIRS is a 23-item scale that assesses broader psychological/interpersonal outcomes associated with erectile dysfunction and its treatment. Each question is rated on a Likert scale from 1 (strongly disagree) to 4 (strongly agree). The scale consists of 3 domains: Sexual Self-Confidence (items 1-6), Spontaneity domain (items 7-15), and Time Concerns (items 16-23). The average domain score for each domain was calculated by adding the nonmissing items for the respective domain, then dividing by the number of nonmissing items for the respective domain. Each average domain score ranged from 1 to 4. Higher scores represent the following: greater sexual self-confidence (better outcome); greater spontaneity (better outcome); higher time concerns (worse outcome). The Least Squares Mean changes were adjusted for treatment group, country, baseline IIEF-EF severity, baseline domain score, and baseline domain score*treatment (if p<0.10).
Time Frame: Baseline, 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline PAIRS observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 252 | 257 | 261
units on a scale
  Sexual Self-Confidence Domain (n=196, 203, 185) | 0.93 [0.83 to 1.03] | 0.90 [0.81 to 1.00] | 0.73 [0.64 to 0.83]
  Spontaneity Domain (n=197, 202, 186) | 0.13 [0.07 to 0.20] | 0.11 [0.04 to 0.18] | 0.02 [-0.05 to 0.09]
  Time Concerns Domain (n=196, 200, 184) | -0.08 [-0.16 to -0.01] | -0.20 [-0.27 to -0.12] | 0.04 [-0.03 to 0.12]

15. Secondary Outcome: Change From Baseline to 4, 8, 16, and 24 Weeks of the Sexual Relationship Domain of the Self-Esteem and Relationship (SEAR) Questionnaire
Description: SEAR assesses psychosocial outcomes in men with erectile dysfunction. Sexual Relationship domain consists of 8 items (items 1-8). Items 2-8 are rated on a scale of 1 (Never) to 5 (Always), whereas item 1 is reverse scored (1=Always and 5=Never). The domain score was computed by summing its respective items, then transforming it into a 0 (least favorable) to 100 (most favorable) scale. Transformed score = 100 x [(actual raw score - lowest possible raw score)/possible raw score range]. Least Squares Mean changes adjusted for baseline score, treatment group, country, visit, and visit*treatment.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline SEAR Sexual Relationship observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 244 | 250 | 246
units on a scale
  Change from Baseline to Week 4 | 27.65 [24.65 to 30.65] | 29.26 [26.29 to 32.23] | 29.50 [26.53 to 32.48]
  Change from Baseline to Week 8 (n=230, 232, 231) | 31.42 [28.23 to 34.61] | 31.07 [27.90 to 34.24] | 31.15 [27.99 to 34.31]
  Change from Baseline to Week 16 (n=167, 146, 101) | 37.59 [34.58 to 40.61] | 32.90 [29.84 to 35.96] | 37.32 [34.03 to 40.60]
  Change from Baseline to Week 24 (n=140, 117, 81) | 39.37 [36.31 to 42.43] | 34.96 [31.79 to 38.13] | 37.46 [34.05 to 40.87]

16. Secondary Outcome: Change From Baseline to 4, 8, 16, and 24 Weeks of the Confidence Domain of the Self-Esteem and Relationship (SEAR) Questionnaire
Description: SEAR assesses psychosocial outcomes in men with erectile dysfunction. Confidence domain measures improvement in confidence; 2 subscales (6 items: Self-Esteem [items 9-12]; Overall Relationship [items 13-14]). Each item range: 1 (Never) to 5 (Always); item 11 reverse scored. Domain score=sum of domain's respective items, then transformed into 0 (least favorable) to 100 (most favorable) scale. Transformed score=100x[(actual raw score-lowest possible raw score)/possible raw score range]. Least Squares Mean change adjusted for baseline score, treatment group, country, visit, and visit*treatment.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline SEAR Confidence observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 245 | 251 | 247
units on a scale
  Change from Baseline to Week 4 | 23.43 [20.32 to 26.54] | 23.04 [19.96 to 26.13] | 25.03 [21.94 to 28.12]
  Change from Baseline to Week 8 (n=230, 233, 232) | 26.97 [23.83 to 30.11] | 26.10 [22.97 to 29.22] | 27.14 [24.03 to 30.25]
  Change from Baseline to Week 16 (n=167, 147, 100) | 33.15 [30.28 to 36.02] | 28.33 [25.41 to 31.25] | 31.86 [28.71 to 35.00]
  Change from Baseline to Week 24 (n=140, 116, 81) | 33.74 [30.64 to 36.84] | 30.42 [27.21 to 33.63] | 31.66 [28.21 to 35.12]

17. Secondary Outcome: Change From Baseline to 4, 8, 16, and 24 Weeks of the Self Esteem Domain of the Self-Esteem and Relationship (SEAR) Questionnaire
Description: SEAR assesses psychosocial outcomes in men with erectile dysfunction. The Self-Esteem domain consists of 4 items (items 9-12), each rated on a scale of 1 (Never) to 5 (Always). Item 11 is reverse scored (1=Always and 5=Never). The domain score was computed by summing its respective items, then transforming it into a 0 (least favorable) to 100 (most favorable) scale. The transformed score = 100 x [(actual raw score - lowest possible raw score)/possible raw score range]. Least Squares Mean changes were adjusted for baseline score, treatment group, country, visit, and visit*treatment.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline SEAR Self-Esteem observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 245 | 251 | 247
units on a scale
  Change from Baseline to 4 Weeks | 25.18 [21.95 to 28.41] | 24.10 [20.90 to 27.30] | 26.59 [23.39 to 29.79]
  Change from Baseline to 8 Weeks (n=230, 233, 233) | 29.14 [25.93 to 32.35] | 27.80 [24.60 to 30.99] | 28.92 [25.75 to 32.10]
  Change from Baseline to 16 Weeks (n=167, 147, 100) | 35.23 [32.20 to 38.26] | 29.46 [26.37 to 32.55] | 33.85 [30.50 to 37.20]
  Change from Baseline to 24 Weeks (n=140, 116, 81) | 35.86 [32.59 to 39.12] | 31.14 [27.75 to 34.52] | 33.52 [29.88 to 37.16]

18. Secondary Outcome: Change From Baseline to 4, 8, 16, and 24 Weeks of the Overall Relationship Domain of the Self-Esteem and Relationship (SEAR) Questionnaire
Description: SEAR assesses psychosocial outcomes in men with erectile dysfunction. The Overall Relationship domain consists of 2 items (items 13-14), each rated on a scale of 1 (Never) to 5 (Always). The domain score was computed by summing its respective items, then transforming it into a 0 (least favorable) to 100 (most favorable) scale. The transformed score = 100 x [(actual raw score - lowest possible raw score)/possible raw score range]. Least Squares Mean changes were adjusted for baseline score, treatment group, country, visit, and visit*treatment.
Time Frame: Baseline, 4, 8, 16, and 24 weeks
Population: The analysis included all randomly assigned participants who had a baseline and post-baseline SEAR Overall Relationship observation.
Measure: Least Squares Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Number analyzed (Participants) | 244 | 251 | 247
units on a scale
  Change from Baseline to Week 4 | 19.92 [16.41 to 23.44] | 21.10 [17.63 to 24.57] | 22.00 [18.52 to 25.48]
  Change from Baseline to Week 8 (n=229, 232, 232) | 22.75 [19.19 to 26.31] | 22.96 [19.43 to 26.50] | 23.74 [20.22 to 27.27]
  Change from Baseline to Week 16 (n=166, 147, 100) | 29.63 [26.46 to 32.79] | 26.96 [23.74 to 30.17] | 28.57 [25.07 to 32.08]
  Change from Baseline to Week 24 (n=139, 116, 81) | 30.28 [26.93 to 33.62] | 29.93 [26.43 to 33.43] | 28.74 [24.93 to 32.56]

ADVERSE EVENTS:
Arm/Group | Tadalafil On Demand | Tadalafil Once a Day | Sildenafil Citrate On Demand
Serious Adverse Events (participants affected / at risk) | 8/250 | 4/257 | 2/260
Other Adverse Events (participants affected / at risk) | 106/250 | 80/257 | 103/260
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil On Demand (N=250) | Tadalafil Once a Day (N=257) | Sildenafil Citrate On Demand (N=260)
Congenital, familial and genetic disorders (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary sequestration (Congenital, familial and genetic disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal disorders (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Pancreatitis acute (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0)
Cholelithiasis (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Hepatobiliary disorders (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
Diverticulitis (Infections and infestations) | 1 (2) | 0 (0) | 0 (0)
Infections and infestations (Infections and infestations) | 2 (3) | 0 (0) | 0 (0)
Parotitis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Metabolism and nutrition disorders (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (5) | 0 (0) | 0 (0)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 1 (5) | 0 (0) | 0 (0)
Colon cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
Neoplasms benign, malignant and unspecified (incl cysts and polyps) (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 (2) | 1 (1) | 1 (2)
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (2)
Completed suicide (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Psychiatric disorders (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
Renal and urinary disorders (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Urinary retention (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Respiratory, thoracic and mediastinal disorders (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Spinal laminectomy (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Surgical and medical procedures (Surgical and medical procedures) | 0 (0) | 1 (1) | 0 (0)
Vascular disorders (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
Venous insufficiency (Vascular disorders) | 1 (2) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tadalafil On Demand (N=250) | Tadalafil Once a Day (N=257) | Sildenafil Citrate On Demand (N=260)
Gastrointestinal disorders (Gastrointestinal disorders) | 21 (52) | 30 (79) | 10 (32)
Infections and infestations (Infections and infestations) | 17 (27) | 10 (22) | 10 (17)
Injury, poisoning and procedural complications (Injury, poisoning and procedural complications) | 44 (117) | 19 (51) | 40 (110)
Intentional overdose (Injury, poisoning and procedural complications) | 16 (40) | 5 (12) | 8 (26)
Overdose (Injury, poisoning and procedural complications) | 21 (56) | 8 (24) | 23 (63)
Musculoskeletal and connective tissue disorders (Musculoskeletal and connective tissue disorders) | 16 (45) | 17 (33) | 9 (20)
Headache (Nervous system disorders) | 10 (30) | 14 (32) | 23 (49)
Nervous system disorders (Nervous system disorders) | 14 (36) | 19 (41) | 27 (60)
Vascular disorders (Vascular disorders) | 11 (37) | 3 (7) | 17 (46)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days